CLINICAL TRIAL: NCT00800787
Title: A Phase 3, Multicenter, Open Label Study to Assess the Safety and Efficacy of Nabi-HB Administered Subcutaneously in Patients With Hepatitis B Virus Associated Liver Disease Who Underwent Liver Transplantation
Brief Title: Nabi-HB Administered Subcutaneously in Patients With Hepatitis B Virus Post Liver Transplantation
Acronym: Nabi-HB-SC
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: New sponsor's existing product under evaluation for this indication
Sponsor: Biotest Pharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4210
Record Dates: First submitted 2008-11-26; First posted 2008-12-02 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2010-06

CONDITIONS: Hepatitis B, Chronic
Keywords: Chronic hepatitis B liver disease
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — hepatitis B hyperimmune globulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm One: Nabi-HB (Experimental): All subjects will be administered Nabi HB Subcutaneously
  Interventions: Biological: Nabi-HB

INTERVENTIONS:
Biological: Nabi-HB — Hepatitis b Immune Globulin (Human)(Nabi-HB) 312 IU/L per dose administered subcutaneously.
  Dosage will be according to each patients body weight, as follow:
  < 75 kg: 500 IU weekly ( may be increase to 1,000 IU weekly if anti-HBs levels are <150 IU/ML > 75 Kg: 1,000 IU weekly
  Other Names: Hepatitis B Immune Globulin (Human)

SUMMARY:
A phase 3, multicenter, open label study to assess the safety and efficacy of Nabi-HB, administered subcutaneously in patients with Hepatitis B Virus Associated Liver Disease who underwent liver transplantation.

DETAILED DESCRIPTION:
This is a phase 3 prospective, single arm open label study to be conducted t approximately 4 study sited located in th e USA. Approximately 25 HBV DNA negative patients who underwent liver transplant at least one year prior, due to chronic hepatitis B infection will bwe eligible for study participation. The study consist of a total of 16 study visit and the duration of participation will be 20 weeks for each patients. Patients will be converted from the intravenous standard HBIG to Nabi-HB subcutaneous administration according to the individual scheduled dosing interval.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years old or older as of visit one.
* If female is not trying to conserve, not lactating, and has a negative serum pregnancy test and use an acceptable method of contraception or be at least one year post-menopausal or surgically sterile.
* Able to provide written informed consent.
* First time liver transplant recipient.
* Primary, single organ recipient (deceased donor <65 years old).
* receive regular long-term HBIG prophylaxis with stabilized HBIG dosage and administration intervals.
* Have negative quantifiable HBV-DNA and HBsAg results prior to dosing at visit 2.
* Following the last IV administration of HBIG, have a baseline serum anti-HBs level of >150 IU/ML prior to dosing at visit 2.

Exclusion Criteria

* Positive HCV or HIV test results.
* Unexplained elevated liver function tests.
* Serum creatinine level >2.0 times the upper limit of normal.
* life expectancy <6 months.
* liver transplantation with ongoing acute rejection episode. Donor liver that was from a hepatitis Bor C positive donor. Underwent a liver transplant <12 months prior to visit 1.
* Know history of cancer, suspected cancer, or cancer therapy within 12 months.
* History of autoimmune disease.
* History/current evidence of coagulation disorder, severe cardiac disease, unhealed gastric or duodenal ulcer, or other significant disease.
* Evidence of any other unresolved infection and any unresolved opportunistic infection requiring treatment.
* Known immunoglobulin A deficiency.
* History of use of immunosupressive or immunomodulatory drug within 3 month prior to visit 1. (except low dose glucocorticoid therapy, <10 mg of prednisone or equivalent per day.)
* received and investigational drug 30 days prior to visit 1.
* use of plasma preparations or other immunoglobulins during the study.
* Know intolerance to proteins of human origin, immunoglobulin, or comparable products.
* Evidence of alcohol and/or drug abuse within 6 month of visit 2 or inability/unwillingness to abstain from alcohol for the duration of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2010-08 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of Nabi-HB administered subcutaneously weekly for a total of 14 weeks in patients who previously underwent a liver transplant. Levels will provide evidence if effective anti-HB levels >150 IU/ML can be maintained. | 14 weeks

SECONDARY OUTCOMES:
To evaluate the safety of Nabi-HB administered subcutaneously weekly for a total of 14 weeks. | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shailesh Chavan, MD, Study Director — Sponsor GmbH